CLINICAL TRIAL: NCT02543125
Title: Nasal High Frequency Oscillatory Versus Nasal Intermittent Positive Pressure Ventilation in Neonate After Extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gao WeiWei (Other)
Responsible Party: Sponsor-Investigator, Gao WeiWei, professor, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: guangdongwchhi4
Record Dates: First submitted 2015-08-21; First posted 2015-09-07 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Insufficiency
Keywords: very low birth weight; respiratory distress; NHFOV; NIPPV
MeSH Terms: conditions — Respiratory Insufficiency; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIPPV (Active Comparator): NIPPV is provided via binasal prongs. Ventilator settings:FiO2:21-40%,peak inspiratory pressure( PIP)：12-22cm H2O,positive and expiratory pressure(PEEP):5-7cm H2O,Rate:30-60 per minute to maintain SaO2 at 90-95%,The weaning process is left to the discretion of the attending physician,when FiO2: 25%,mean airway pressure (MAP)<6cm H2O,R:30 per minute .
  Interventions: Device: NIPPV
- NHFOV (Active Comparator): NHFOV is provided via binasal prongs. Ventilator settings:FiO2:21-40%,MAP：6-14 cm H2O,Hertz(HZ):5-10 to maintain SaO2 at 90-95%,The weaning process is left to the discretion of the attending physician,when FiO2: 25%,mean airway pressure (MAP)<6cm H2O.
  Interventions: Device: NHFOV

INTERVENTIONS:
Device: NIPPV — For infants in the NIPPV-group who "fail"NIPPV (see definition below), need immediate intubation, a invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  Other Names: SLE 5000
  Arms: NIPPV
Device: NHFOV — For infants in the NHFOV-group who "fail"NHFOV (see definition below), need immediate intubation, a invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  Other Names: SLE 5000
  Arms: NHFOV

SUMMARY:
To evaluate the efficacy and safety of nasal high frequency oscillatory ventilation(NHFOV) in preterms with respiratory disease syndrome(RDS) after extubation.

DETAILED DESCRIPTION:
To very low birth weight infant(VLBW) with respiratory disease syndrome(RDS) who need mechanical ventilation,early extubation may have more benefits.Early extubation may decrease the ventilation-associated pneumonia(VAP),sepsis and decrease the incidence of severity bronchopulmonary dysplasia(BPD).But often fail attempts at extubation because of apnea,atelectasis,hypercapnia,hypoventilation or other illnesses.

High frequency oscillatory ventilation is benefit to lung.Initial ventilation with HFOV in preterm with RDS may reduce the incidence of BPD and improve the neurodevelopment.Compared HFOV with conventional ventilation in preterm infants showed that HFOV had superior lung function when 11 to 14 years age.Whether nasal high frequency oscillatory ventilation(NHFOV) also have those advantages in non-invasive mode? Null D M et al do a experiment on preterm lambs,the result suggest that NHFOV may promotes alveolarization.But there was no clinical trials to prove.

The nasal intermittent positive pressure ventilation (NIPPV) group fail definition：1、 Fraction of inspired oxygen (FiO2)>40%、MAP>12 centimeter water column (cm H2O),but arterial oxygen saturation (SaO2)<90%.2、significant abdominal distension.3、PaCO2>60millimeter of mercury(mmHg)or partial pressure of arterial oxygen (PaO2)<45 millimeter of mercury(mmHg).4、severe apnea( definition:>6 episodes requiring stimulation in 6 hours or requiring >1 episodes of positive-pressure ventilation) 5.potential of hydrogen (PH)<7.2 The

The NHFOV group fail definition：1、FiO2>40%、MAP>14 mbar,but SaO2<90%.2、significant abdominal distension.3、PaCO2>60millimeter of mercury(mmHg) or PaO2<45millimeter of mercury(mmHg).4、severe apnea 5.PH<7.2.

ELIGIBILITY:
Inclusion Criteria:

1. birth weight>1000g
2. gestational age >28 weeks
3. have respiratory distress syndrome and need invasive ventilation

Exclusion Criteria:

1. birth wight<1000g
2. gestational age <28 weeks
3. infants wiht abnormalities of upper and lower airways
4. infants have contraindications of non-invasive ventilation -

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
intubation rate | 72 hours
  endotracheal intubation rate assessed within 72 hours after extubation

SECONDARY OUTCOMES:
significant apnea | 7 days
  significant apnea measured by Colin J definition:6 episodes requiring stimulation in 6 hours or requiring > 1episodes of positive ventilation
air leaks | 3 months
  air leaks assessed by chest X-ray
Bronchopulmonary dysplasia | 3 months
  Bronchopulmonary dysplasia assessed by national institute of child health and human development definition
necrotizing enterocolitis | 3 months
  necrotizing enterocolitis assessed by abdominal X-ray and Bell classification

CONTACTS AND LOCATIONS:
Overall Officials: yang jie, doctor, Study Director — Guangdong Women and Children Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Donn SM, Sinha SK. Minimising ventilator induced lung injury in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F226-30. doi: 10.1136/adc.2005.082271. PMID 16632652
- [Result] van der Hoeven M, Brouwer E, Blanco CE. Nasal high frequency ventilation in neonates with moderate respiratory insufficiency. Arch Dis Child Fetal Neonatal Ed. 1998 Jul;79(1):F61-3. doi: 10.1136/fn.79.1.f61. PMID 9797628
- [Result] Colaizy TT, Younis UM, Bell EF, Klein JM. Nasal high-frequency ventilation for premature infants. Acta Paediatr. 2008 Nov;97(11):1518-22. doi: 10.1111/j.1651-2227.2008.00900.x. Epub 2008 Jun 9. PMID 18549418
- [Result] De Luca D, Carnielli VP, Conti G, Piastra M. Noninvasive high frequency oscillatory ventilation through nasal prongs: bench evaluation of efficacy and mechanics. Intensive Care Med. 2010 Dec;36(12):2094-100. doi: 10.1007/s00134-010-2054-7. Epub 2010 Sep 21. PMID 20857278
- [Result] Null DM, Alvord J, Leavitt W, Wint A, Dahl MJ, Presson AP, Lane RH, DiGeronimo RJ, Yoder BA, Albertine KH. High-frequency nasal ventilation for 21 d maintains gas exchange with lower respiratory pressures and promotes alveolarization in preterm lambs. Pediatr Res. 2014 Apr;75(4):507-16. doi: 10.1038/pr.2013.254. Epub 2013 Dec 30. PMID 24378898
- [Result] Fischer HS, Bohlin K, Buhrer C, Schmalisch G, Cremer M, Reiss I, Czernik C. Nasal high-frequency oscillation ventilation in neonates: a survey in five European countries. Eur J Pediatr. 2015 Apr;174(4):465-71. doi: 10.1007/s00431-014-2419-y. Epub 2014 Sep 18. PMID 25227281